CLINICAL TRIAL: NCT01100463
Title: A Phase 1-2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Pharmacokinetic Profile of 0.1% Uracil Topical Cream (UTC) in the Prevention of Hand-Foot Syndrome (HFS) in Patients With Metastatic Breast Cancer Treated With Capecitabine
Brief Title: Study of 0.1% Uracil Topical Cream (UTC) for the Prevention of Hand-Foot Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanometics (d.b.a. PHD Biosciences) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OIC-1UO-C001
Record Dates: First submitted 2010-04-06; First posted 2010-04-09 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Palmar-Plantar Erythrodysesthesia; Breast Cancer
Keywords: HFS, Hand-Foot Syndrome, Capecitabine, Breast Cancer
MeSH Terms: conditions — Hand-Foot Syndrome; Breast Neoplasms; Hyaline Fibromatosis Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Lotion (Placebo Comparator)
  Interventions: Drug: Cream
- 0.1% Uracil (Experimental)
  Interventions: Drug: 0.1% Uracil Cream

INTERVENTIONS:
Drug: Cream — Twice daily lotion to prevent HFS
  Arms: Placebo Lotion
Drug: 0.1% Uracil Cream — Twice daily lotion to prevent HFS
  Arms: 0.1% Uracil

SUMMARY:
The purpose of this research study is to see if combining uracil cream (UTC) with capecitabine (Xeloda) can prevent Hand-Foot Syndrome. The study will also see what effects UTC and capecitabine may have in patients with metastatic breast cancer.

DETAILED DESCRIPTION:
Capecitabine is used in the treatment of human breast cancer among other human cancers. Following absorption, capecitabine is converted enzymatically to 5-fluorouracil (5-FU). The administration of capecitabine or 5-FU can cause a cutaneous toxicity known as hand-foot syndrome (HFS) or palmar-plantar erythrodysesthesia (PPE). HFS is progressive with dose and duration of exposure to 5-FU or capecitabine. HFS is characterized by progressive redness and cracking of hands and feet. Currently, there are no approved therapies for HFS.

ELIGIBILITY:
Inclusion Criteria:

* Females, at least 18 years old
* Histologically or cytologically confirmed metastatic breast cancer
* You also cannot have any ulcerations or open wounds on palms of hands or soles of feet

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C)prior to entering the study or if you have not recovered to Grade 1 or better (except for alopecia)from adverse events due to agents administered more than 2 weeks earlier.
* Use vitamin 6, chronic use of Cox-2 inhibitors, use full-dose anti- coagulants or use nicotine patches.

The above is not a complete list of eligibility criteria. Please see your study doctor for more information.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Grade 2 and 3 HFS as graded by Roche Criteria | Maximum of 6 months of therapy
  * Time to first HFS event
  * Requirements for capecitabine dose reduction/interruption due to HFS
  * Digital Photos will be taken of the hands and feet at specific intervals
Serum Pharmacokinetic Levels of Uracil will be drawn | Maximum of 6 months of therapy
  Pharmacokinetic levels will be drawn at specific intervals

SECONDARY OUTCOMES:
Anti-Tumor efficacy of Capecitabine | Maximum of 6 months of therapy
  RECIST - Radiologic Criteria for subjects with measurable disease

CONTACTS AND LOCATIONS:
Overall Officials: James Cantrell, MD, Principal Investigator — Birmingham Hematology/Oncology Associates
Locations (6):
- United States (6):
  - Bruno Cancer Center, Birmingham, Alabama
  - Comprehensive Cancer Center, Palm Springs, California
  - Research Institute of Deaconess Clinic, Evansville, Indiana
  - Cancer Care Center, New Albany, Indiana
  - Kansas City Cancer Centers, Overland Park, Kansas
  - Signal Point Clinical Research Center, Middleton, Ohio